CLINICAL TRIAL: NCT04608006
Title: Epidural Analgesia and Delivery of Second Twin: Prospective Observational Study
Brief Title: Epidural Analgesia and Delivery of Second Twin
Acronym: Epidural
Status: Completed | Type: Observational
Sponsor: Abdelrady S Ibrahim, MD (Other)
Responsible Party: Sponsor-Investigator, Abdelrady S Ibrahim, MD, Assiut University Faculty of Medicine Anesthesia Dept, Assiut University
Organization: Assiut University (Other)
Other Study IDs: IRB0000871247; Assiut Universitr (Other: Faculty of Medicine); Ain Shams University (Other: Faculty of Medicine)
Record Dates: First submitted 2020-10-23; First posted 2020-10-29 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Epidural; Analgesia; Labor Pain
Keywords: Epidural; Analgesia; Labour
MeSH Terms: conditions — Agnosia; Labor Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Vaginal Delivery: Delivered both twins vaginally
  Interventions: Drug: Bupivacaine-fentanyl
- C-Section Delivery: Delivered both twins by Cesarean Section
  Interventions: Drug: Bupivacaine-fentanyl
- Vaginal/C-Section Delivery: Delivery first twin vaginally and second twin By C-Section.
  Interventions: Drug: Bupivacaine-fentanyl

INTERVENTIONS:
Drug: Bupivacaine-fentanyl — Initial epidural bolus of 10 ml Bupivacaine 0.125% plus 50 mcg Fentanyl, followed by continuous infusion pf Bupivacaine 0.0625%™ plus 1mcg/dl Fentanyl
  Other Names: Epidural Catheter insertion

SUMMARY:
Over an 8-year period, 124 twin pregnancies at gestational age ≥32 weeks with both twins presenting as a vertex and eligible for vaginal delivery were reviewed. Excluded were patients with the following intrapartum factors which may affect mode of delivery of second twin: 1. Presentation of the 2nd twin: breech or other than vertex; 2. Monochorionic twins; 3. Induction of labour; 4. difference in foetal weight between twin B and twin A ≥25%. The chi-square statistic was used to compare differences in the incidence of retained second twin between the groups.

DETAILED DESCRIPTION:
The investigators conducted this prospective study in women with twins pregnancy planned for trial of vaginal delivery and gave birth between January 2014 and December 2019, in the Department of obstetrics and Gynaecology of the Sabah Maternity Hospital, Sabah Specialized Area, Kuwait. The Sabah Maternity Hospital is a tertiary care hospital for the country of Kuwait with approximately 12500 deliveries per year. The study protocol was approved by the Ethics Committee.

ELIGIBILITY:
Inclusion Criteria:

.gestational age of 32 weeks, determined by an early ultrasound performed in the second trimester or certain last menstrual period; (2) both twins viable; (3) eligibility for vaginal delivery as defined by twin A being cephalic; and (4) no previous cesarean section.

Exclusion Criteria:

* underwent an elective or repeat cesarean section
* presentation of twin B at delivery other than cephalic (breech, oblique or transverse presentation
* induction of labour
* the difference in foetal weight between twin B and twin A at delivery ≥25% .Neonates were excluded if one was stillborn or had major congenital malformations.

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Study Population: Women with twins pregnancy planned for trial of vaginal delivery and gave birth
Sampling Method: Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2014-11-03 (Actual); Primary Completion 2019-12-24 (Actual); Study Completion 2019-12-24 (Actual)

PRIMARY OUTCOMES:
Delivery of First twin | 24 hours
  Vaginal or C-Section
Delivery of Second twin | 24 hours
  C-Section or C-Section

CONTACTS AND LOCATIONS:
Overall Officials: Abdelrady S Ibrahim, M.D., Principal Investigator — Assiut University
Locations (1):
- Assiut university faculty of medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Alexander JM, Sharma SK, McIntire DD, Leveno KJ. Epidural analgesia lengthens the Friedman active phase of labor. Obstet Gynecol. 2002 Jul;100(1):46-50. doi: 10.1016/s0029-7844(02)02009-4. PMID 12100802